CLINICAL TRIAL: NCT04766905
Title: Mini Lateral Shoulder Approach
Acronym: MLSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Issa, Abdulhamid Sayed, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Second Sayed Issa's Approach
Record Dates: First submitted 2021-02-12; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Shoulder Impingement Syndrome; Rotator Cuff Tendinopathy; Adhesive Capsulitis and Frozen Shoulder Syndrome
Keywords: Shoulder; Shoulder approach; Lateral Shoulder approach; Shoulder impingement syndrome; Rotator cuff tendinopathy; Adhesive capsulitis; Frozen shoulder syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome; Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Issa1 (Experimental): Dr.A.Sayed Issa and his team
  Interventions: Procedure: Mini Lateral Shoulder Approach (MLSA)

INTERVENTIONS:
Procedure: Mini Lateral Shoulder Approach (MLSA) — The skin incision is about 4 to 5 cm made by the distal acromial edge in sagittal plane, The dissection takes place slightly over the acromial edge proximally and over the origin of the acromial deltoid part (the middle part of deltoid origin) distally.
  After clearly revealing the region of the medial deltoid origin on the acromion, the acromionic deltoid origin is skinned only; of the edge of the acromion, and that maybe accrued by electric knife pen or periosteal elevator, without exposure the clavicular deltoid origin in the front and the deltoid origin on the spine of scapula in the back, the origin of the acromial deltoid is distanced laterally and distally, where the lateral edge, the lower surface of the acromion, under acromial bursa and the rotator cuff are exposed clearly.
  Other Names: Second Sayed Issa's Approach

SUMMARY:
The incision is very useful and easy for the direct lateral shoulder joint exposure.

DETAILED DESCRIPTION:
The skin incision is about 4 to 5 cm made by the distal acromial edge in sagittal plane, The dissection takes place slightly over the acromial edge proximally and over the origin of the acromial deltoid part (the middle part of deltoid origin) distally.

After clearly revealing the region of the medial deltoid origin on the acromion, the acromionic deltoid origin is skinned only; of the edge of the acromion, and that maybe accrued by electric knife pen or periosteal elevator, without exposure the clavicular deltoid origin in the front and the deltoid origin on the spine of scapula in the back, the origin of the acromial deltoid is distanced laterally and distally, where the lateral edge, the lower surface of the acromion, under acromial bursa and the rotator cuff are exposed clearly.

Throw this approach can be made acromioplasty and rotator cuff tears repair especially upper part of rotator cuff tear very easily.

For wound closure the acromionic deltoid origin is reattached to the acromial edge by long period synthetic absorbable sutures as PDS and PDO, or non absorbable sutures as Polyester suture, under skin and skin sutures are made.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented with Shoulder Impingement Syndrome refractory to conservative treatment and local steroid injection
* Patients presented with Adhesive Capsulitis and Frozen Shoulder Syndrome refractory to conservative treatment and local steroid injection
* Patients without femur head immigration on X-ray
* Patients with injury for one month to six months maximum

Exclusion Criteria:

* Patients with femur head immigration on X-ray
* Patients with injury for more than six months
* Un controlled diabetes mellitus type 1 and 2
* Patients with non controlled Vascular hypertension
* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
* Myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization
* Patients with history of Carpal Tunnel release surgery failure

Ages: 16 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2021-01-17 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
Less surgical procedure time than traditional approaches | up to two years
  25 minutes to 45 minutes, it's depends of rotator cuff tear if exist or not.
Less rehabilitation time than traditional approaches | up to two years
  6 - 8 weeks
Passive physiotherapy immediately | up to two years
  next day of surgery
Active physiotherapy without rotator cuff tear | up to two years
  after two weeks of surgery
Mini cosmetic incision to the shoulder | up to two years
  4 - 5 cm
Active physiotherapy with rotator cuff tear | up to two years
  after three weeks of surgery

SECONDARY OUTCOMES:
very good patients satisfaction | up to two years
  after 8 weeks
Restore deltoid muscle strength | up to two years
  about 3 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Sayed Issa's Clinic, Aleppo, Syria